CLINICAL TRIAL: NCT05569889
Title: Impact of Implementing of Custom Surgical Tray (CST) in Anterior Cruciate Ligament Reconstruction Procedure on Sustainable Development.
Brief Title: Custom Surgical Tray in ACLR Procedure
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RnIPH 2021-104
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Custom Surgical Tray; Sustainable Development
MeSH Terms: interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: The medical staff was using the traditional surgical draping kit and single-packed sterile instruments (SPSI) that have to be opened separately
  Interventions: Procedure: Anterior Cruciate Ligament reconstruction (ACLR)
- experimental group: The medical staff was using only the single packed CST, and containing all the necessary single-use items like surgical blades, sutures, dressing, surgical drapes, syringes, compresses, surgical gloves, jerseys.
  Interventions: Procedure: Anterior Cruciate Ligament reconstruction (ACLR)

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament reconstruction (ACLR) — A comparison between the two groups were done regarding the three following stages: (a) the preparation time of the trolley, which is the time taken by the CNOR to recover from the reserves all the single-packed sterile instruments (SPSI) necessary for the intervention or to recover the CST (b) the opening time of the instruments by the circulating nurse who opens the packages and gives them to the surgical nurse while respecting the sterility of the items, and by the surgical nurse who prepares the table for the intervention, and (c) the sorting time of the waste between plastic and paper at the end of the intervention.

SUMMARY:
In the Toulouse University Hospital, the Custom Surgical Tray (CST) were not referenced. The nurse had to prepare and open all the components of the procedure separately. This is a long and wasteful process.

CST brings together all the single-use medical devices necessary for an intervention, including draping and dressing elements, in the same single packaging.

Following the new local call for tenders on draping kits, and with the aim of standardizing and rationalizing practices, the implementation of CST within the requesting blocks whose orthopedic and traumatology block has been validated.

The hypothesis is that the CST would save time on preparing the trolley and on opening single-use equipment in the room while limiting the amount of waste.

DETAILED DESCRIPTION:
To determine the social impact, the study assess the quality of life at work by measuring the difference, after implementing CST, in time needed for preparation of the trolley before entering the OR, for opening the instruments necessary by the surgical and circulating certified perioperative nurse (CNOR) in the Operating Room (OR), and for sorting the waste derived from the instrument's packages between plastic and paper after the intervention. In addition, the study assessed the biomechanical risk factors related to musculoskeletal disorders by evaluating the number of movements made by the CNOR when opening the instruments and sorting the waste, with and without CST. Finally, the study evaluate CNOR and surgeon's satisfaction after the implementation of CST.

To determine the ecologic impact, the difference in the number and weight of waste due to packaging of the disposable instruments, with and without CST was evaluated.

To determine the economic impact, the difference in cost of the instruments used, with and without CST was evaluated.

The hypothesis is that the use of CST enhances Sustainable Development (SD) by maintaining social development and environment protection, despite a possible additional cost.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old patients
* patient necessitating a Anterior Cruciate Ligament reconstruction

Exclusion Criteria:

* patient refusing to participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All surgery of Anterior Cruciate Ligament reconstruction were study during the period between 15 february 2021 and 15 August 2021.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Preparation time of the trolley | 1 day
  Compared the number of minutes to prepare the trolley between control and experimental group
Opening time of the instruments | 1 day
  Compared the number of minutes to open all the instrument between control and experimental group
Sorting time of the waste | 1 day
  Compared the number of minutes to sorting of the waste between control and experimental group

SECONDARY OUTCOMES:
weight of trash packages | 1 day
  Compared the weight in grams of trash packages between control and experimental group
Number of TRASH packages | 1 day
  Compared the Number of trash packages between control and experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CAVAIGNAC, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No